CLINICAL TRIAL: NCT02529800
Title: A Randomized, Open-label, Single Dose, Three-way Crossover Clinical Trial to Investigate the Pharmacokinetics Incorporating a Comparison of Fed/Fasted Pharmacokinetics of HIP1402 in Healthy Male Volunteers
Brief Title: Investigating the Pharmacokinetic Characteristics of HIP1402 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-VICT-102
Record Dates: First submitted 2015-08-13; First posted 2015-08-20 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sequence 1 (Experimental): High fat diet+HGP0412 → High fat diet+HIP1402 → fasted state+HIP1402
  Interventions: Drug: HIP1402; Drug: HGP0412
- Sequence 2 (Experimental): High fat diet+HIP1402 → fasted state+HIP1402 → High fat diet+HGP0412
  Interventions: Drug: HIP1402; Drug: HGP0412
- Sequence 3 (Experimental): fasted state+HIP1402 → High fat diet+HGP0412 → High fat diet+HIP1402
  Interventions: Drug: HIP1402; Drug: HGP0412

INTERVENTIONS:
Drug: HIP1402 — Tamsulosin HCl 0.4mg
Drug: HGP0412 — Tamsulosin HCl 0.2mg

SUMMARY:
To investigate the PK charateristics and the effect of food on the PK in healthy male volunteers who receive HIP1402 capsule in fed versus fasted condition

DETAILED DESCRIPTION:
A randomized, open-label, single dose, three-way crossover clinical trial to investigate the pharmacokinetics incorporating a comparison of fed/fasted pharmacokinetics of HIP1402 in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteer, age 19~50 years
2. Weight ≥55kg and ≤90kg, The result of Body Mass Index(BMI) is not less than 18 kg/m2 , no more than 27 kg/m2
3. Subject who has the ability to comprehend the study objectives, contents and the property of the study drug before participating in the trial
4. Subject who has the ability and willingness to participate the whole period of trial

Exclusion Criteria:

1. Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in kidney, liver, cardiovascular system, respiratory system, endocrine system, or neuropsychiatric system.
2. History of relevant drug allergies or clinically significant hypersensitivity reaction.
3. Systolic Blood Pressure: lower than 100mmHg or higher than 150mmHg, Diastolic Blood Pressure: lower than 60mmHg or higher than 100mmHg
4. Liver enzyme (AST, ALT) level exceeds the maximum normal range more than one and a half times.
5. Subjects who took prescription drugs within 14 days from the patient screening or non-prescription medicine within 7 days which can affect the result of this clinical trial (acceptable according to the investigator's judgement)
6. Intake of more than 210g of alcohol per week or who can't abstain from alcohol during the trial.
7. Subjects who smoke more than 10 cigarettes per day or who can't quit smoking during the trial.
8. Positive screening on Hepatitis B surface antigen(HBsAg), anti-Hepatitis C virus(HCV) or anti-Human immunodeficiency virus(HIV).
9. Subjects who judged ineligible by the investigator.

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Tamsulosin, AUC(AUClast, AUCinf), | pre-dose(0 h), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 h post-dose
Tamsulosin, Cmax | pre-dose(0 h), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 h post-dose
Tamsulosin, Tmax | pre-dose(0 h), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 h post-dose
Tamsulosin, t1/2 | pre-dose(0 h), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 h post-dose
Tamsulosin, CL/F | pre-dose(0 h), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 h post-dose
Tamsulosin, Vz/F | pre-dose(0 h), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 h post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, M.D., Principal Investigator — Seoul National University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ban MS, Kim YK, Kim B, Jung J, Kim YI, Oh J, Yu KS. Evaluation of the pharmacokinetics and food effects of a novel formulation tamsulosin 0.4 mg capsule compared with a 0.2 mg capsule in healthy male volunteers. Transl Clin Pharmacol. 2020 Dec;28(4):181-188. doi: 10.12793/tcp.2020.28.e17. Epub 2020 Nov 24. PMID 33425801